CLINICAL TRIAL: NCT02772536
Title: An Open Design Clinical Trial Investigating the Effect of Tinted Light on Perception of Tinnitus to Establish Its Efficacy
Brief Title: A Clinical Trial Investigating Effect of Tinted Light on Perception of Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: Leicester Royal Infirmary NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0473
Record Dates: First submitted 2016-05-04; First posted 2016-05-13 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Tinnitus
Keywords: Chronic Tinnitus Tinted Light Change in Perception
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Visual Stimulus Condition Set (Other): In this single arm study all participants are subject to a set of three visual stimulus conditions.
  These are: Low ambient light; Self selected tinted light; White light
  Interventions: Other: Visual Stimulus Condition Set

INTERVENTIONS:
Other: Visual Stimulus Condition Set — In this single arm study, all participants are subject to a set of three visual stimulus conditions.
  Low ambient light for 10 mins: Self selected tinted light (20 Mins); White light (20 mins).
  VAS/CGI scores for each stimulus condition in the above set are reported at five minute intervals.

SUMMARY:
Background

An earlier pilot study provided evidence that about 40% of tinnitus sufferers reported that viewing particular tints of light appeared to result in some improvement of their tinnitus.

This ameliorative effect appeared to be primarily acute and only reported to occur whilst viewing the tint. Individual patients would choose differing tints with some identifying more than one tint that affected their tinnitus.

Aim of the Study

In this current basic science study, the aim is to provide preliminary data to return estimates of the efficacy of using tinted light to ameliorate tinnitus.

After identification of responders during screening, responders are invited to attend three further trial sessions, where their tinnitus is assessed in response to three luminance conditions: Low Ambient Light; Tint of Light affecting Tinnitus; White Light.

The response to low ambient light serves as a control to compare the effect of tinted light against and the response to white light serves as an 'active' stimulus comparator.

These results will then establish whether tinted light provides patients with a useful improvement in their tinnitus compared with measures of their baseline tinnitus obtained in the dark and against a standardised white light stimulus.

They will also inform further development of the technique as a potential treatment for tinnitus in responsive patients.

Over the three sessions, the averaged responses given by the patient under each stimulus condition will be analysed to provide a measure of efficacy.

DETAILED DESCRIPTION:
Study Protocol

The overall study design is open, as participants are explicitly required to identify a specific light tint that they perceive as affecting the annoyance or intrusiveness of their tinnitus. An element of an active control is provided by reference to changes reported with a self-selected tint referenced against white light. The a priori assumption is that with this optically defined white light, the reported changes in tinnitus will remain as zero. The following is a protocol outline of the trial as experienced by participants. All trial data is anonymised with hard copies securely held at the trial site.

Invitation to participate and seeking consent

First Visit:

Questionnaires and Screening for identifying Tinnitus patients reporting their whose perception of tinnitus is changed by tinted light .

Trial Questionnaires Following consent to take part in the study, at the first visit the participant completes two questionnaires. This provides relevant baseline demographics, history of general health tinnitus and hearing. The second questionnaire is the Oregon Tinnitus Functional Index (TFI) to assess the impact of tinnitus on the participant's life.

Light Test Screening:

Identification of Tints Affecting Tinnitus Perception The following all take place in a sound proof room at the Leicester Royal Infirmary in which the participant is comfortably seated during the session.

After an explanation of what will be asked of them, the patient is asked to provide Tinnitus Annoyance and Tinnitus Loudness VAS values to serve as baseline measurements.

The only sources of illumination during the experimental procedure are from the Light Emitting Diode (LED) lamp in front of the patient and indirect low level ambient illumination from a laptop screen. The laptop screen is viewed by the experimenter and its display cannot be seen by the participant.

The LED lamp consists of three banks of Red, Green and Blue (RGB) LEDs under direct manual and computer control. The Lamp head projects down onto an A4 sized platen that forms the base of the lamp. On this platen base, an A4 sheet of white paper is illuminated by the calibrated output of the RGB LED.

The participant is then comfortably seated and asked to look at the default setting of white illuminated by the calibrated LED lamp. This is at a distance of about 45-50 cm. The participant then controls the colour output of the LED lamp by varying three independent manual dials, one each for the Red, Green and Blue LEDs to produce a very wide range of light tints. A demonstration and practice with explanation by the experimenter is provided prior to commencing this procedure.

During the screening procedure, the patient is asked to report if any of the tints they see appears to improve their tinnitus. The individual RGB values for each tint reported by the participant are recorded by the experimenter.

The degree of improvement is estimated by the patient reporting Tinnitus Annoyance and Loudness VAS ratings as described below and a Clinical Global Index (CGI) value as described below.

If they do identify one or more tinnitus ameliorating tints, then they are invited to replicate this again and the settings return to the default optical white. The RGB dials do not have any calibration marking, but are connected to a laptop that monitors the colour space generated.

This is under experimenter control. The individual RGB values for each tint reported by the participant are again recorded by the experimenter along with the two Tinnitus VAS and a CGI value.

The experimenter also establishes if the chosen tint can be replicated independently under computer control by gradually changing the RGB values to replicate the tint(s) along with the recording of VAS and CGI values as described above.

Importantly, no verbal feedback by the experimenter about tint choice is given and the only guide assumed to be active in tint choice is effect on the participants tinnitus.

Once replication has been established at the first screening session the participant is then invited to attend a further three sessions to provide evidence of stability of longer term effect necessary to demonstrate efficacy.

Second to Fourth Visit: Estimating Efficacy On these visits, the participant is invited back into the soundproof room and is seated comfortably in front of the LED lamp.

At the start of the second session, patients are asked to provide their baseline VAS ratings for tinnitus loudness and annoyance. At this second visit, the patient is then invited to choose what they consider to be their optimal tint fro improving their tinnitus as they did at the first visit.

The optimal tint affecting their tinnitus is then replicated by both the patient and independently by the experimenter.

Once they have confirmed their optimal choice, the setting is noted by the experimenter for presentation.

The patient is then presented with three sets of visual stimulus condition to assess efficacy.

Low level ambient lighting: - Under low level illumination patients will be asked to provide VAS and CGI ratings for their tinnitus on three occasions over 10 minutes at 0,5 and 10 mins. These values are recorded by the experimenter.

Optimal tint - Patients will view their optimal light tint presented for 20 minutes and asked to provide VAS and CGI ratings on three occasions at 5, 10 and 15 mins. At 0 and 20 mins, i.e. just before and just after the optimal tint is presented, they are asked to provide these values under conditions of low ambient illumination. These values are recorded by the experimenter.

White Light - After a few minutes interval, patients are asked to repeat the above procedure but whilst viewing white light that serves as an active comparator. These values are recorded by the experimenter.

The third and fourth visits are ideally spaced at two weekly intervals, but timings of the visits are arranged to fit with the lifestyle and commitments of the patients.

At these visits, the patients are again invited to provide VAS and CGI scores to the three illumination conditions described above.

Once a full set of data from the four visits has been obtained, the patient has completed their participation in the trial. The VAS and CGI measurements obtained are then further processed to return primary and secondary outcome measures for each patient at the end of their participation in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 + years
* Not receiving other tinnitus therapy or involved in any other tinnitus trial
* To be in reasonable or good general health
* Willing and able to give informed consent for participation in the study
* Able to understand simple verbal explanation in English
* Able to provide simple clear verbal feedback in English

Exclusion Criteria:

* Aged under 18 yrs
* Suffering only acute occasional tinnitus or non-intrusive tinnitus
* Any serious illness that may adversely affect participation for example cancer, dementia/neurodegenerative illness, psychoses, stroke
* Receiving other treatments for tinnitus during the trial
* Unable or unwilling to give consent
* Unable to understand or speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-03-10 (Actual); Primary Completion 2017-12-09 (Actual); Study Completion 2017-12-09 (Actual)

PRIMARY OUTCOMES:
Averaged difference between dark and optimal tint tinnitus annoyance Visual Analogue Score (VAS) | At the end of the participation period in the efficacy phase of trial, typically 4-6 weeks.
  As described in the protocol, during the efficacy phase of the trial, the participant attends clinic on three occasions. At each visit, the participant provides tinnitus annoyance VAS values at set time points during the presentation of the three visual stimulus conditions (dark, optimal light tint, white light). At the end of each visit, the tinnitus annoyance VAS for the different visual stimulus conditions is then averaged. The difference between the averaged annoyance VAS for dark and the optimal light tint is calculated for each visit.
  After the final visit, the difference between the dark and optimal light tint conditions over all three visits is then averaged. This averaged difference in tinnitus annoyance over all three visits is then used as the primary outcome measure for the study.

SECONDARY OUTCOMES:
Averaged difference between dark and optimal tint tinnitus loudness Visual Analogue Score (VAS) | At the end of the participation period in the efficacy phase of trial, typically 4-6 weeks.
  As described in the protocol, during the efficacy phase of the trial, the participant attends clinic on three occasions. At each visit, the participant provides tinnitus loudness VAS values at set time points during the presentation of the three visual stimulus conditions (dark, optimal light tint, white light).
  At the end of each visit, the tinnitus loudness VAS for the different visual stimulus conditions is then averaged. The difference between the averaged loudness VAS for dark and the optimal light tint is calculated for each visit.
  After the final visit, the difference between the dark and optimal light tint conditions over all three visits is then averaged. This averaged difference in tinnitus loudness over all three visits is then used as a secondary outcome measure for the study.

OTHER OUTCOMES:
Averaged difference between dark and optimal tint Clinical Global Index Values | At the end of the participation period in efficacy phase of trial, typically 4-6 weeks.
  As described in the protocol, during the efficacy phase of the trial, the participant attends clinic on three occasions. At each visit, the participant provides CGI values at set time points during the presentation of the three visual stimulus conditions (dark, optimal light tint, white light).
  At the end of each visit, the CGI values for the different visual stimulus conditions are then averaged. The difference between the averaged CGI value dark and the optimal light tint is calculated for each visit.
  After the final visit, the difference in CGI values over the dark and optimal light tint conditions over all three visits is then averaged. This averaged CGI value difference over all three visits is then used as a further secondary outcome measure for the study.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mulheran, PhD, Study Director — University of Leicester
Locations (1):
- Leicester Royal Infirmary University Hospitals Trust, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No